CLINICAL TRIAL: NCT00670358
Title: Phase I/II Study of Lenalidomide (Revlimid), Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone (R2CHOP) Chemoimmunotherapy in Patients With Newly Diagnosed Diffuse Large Cell and Follicular Grade IIIA/B B Cell Lymphoma
Brief Title: Lenalidomide, Rituximab, and Combination Chemotherapy in Treating Patients With Newly Diagnosed Stage II, Stage III, or Stage IV Diffuse Large Cell or Follicular B-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC078E; MC078E (Other: Mayo Clinic Cancer Center); RV-NHL-PI-0325 (Other: Celgene Protocol); 07-007992 (Other: Mayo Clinic IRB); NCI-2009-01196 (Registry Identifier: NCI CTRP); P50CA097274 (NIH)
Record Dates: First submitted 2008-04-30; First posted 2008-05-01 (Estimated); Results first posted 2022-11-17 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — pegfilgrastim; Rituximab; Cyclophosphamide; Doxorubicin; Lenalidomide; Prednisone; Vincristine; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: pegfilgrastim
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: lenalidomide
Drug: prednisone
Drug: vincristine sulfate
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Lenalidomide may stimulate the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with rituximab and combination chemotherapy may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of lenalidomide when given together with rituximab and combination chemotherapy and to see how well they work in treating patients with newly diagnosed stage II, stage III, or stage IV diffuse large cell or follicular B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of lenalidomide when given in combination with rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone in patients with newly diagnosed stage II-IV diffuse large cell or grade 3 follicular B-cell lymphoma. (Phase I)
* To assess the efficacy of this regimen, in terms of event-free survival and response rate, in these patients. (Phase II)
* To assess the safety of this regimen in these patients. (Phase II)

Secondary

* To assess the host immune function at baseline and after treatment and correlate these parameters with tumor response and event-free survival.

OUTLINE: This is a multicenter, phase I dose-escalation study of lenalidomide followed by a phase II study.

* Phase I: Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1, oral prednisone on days 1-5, and oral lenalidomide on days 1-10. Patients also receive pegfilgrastim subcutaneously on day 2. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients receive lenalidomide at the maximum tolerated dose determined in phase I and rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine, prednisone, and pegfilgrastim as in phase I.

Blood is collected at baseline, before course 3, and after completion of study treatment for translational research studies. Research studies include immune function and cytokine analysis, T- and B- quantitative lymphocyte analysis, and single nucleotide polymorphism analysis.

After completion of study therapy, patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large cell or grade 3A/B follicular lymphoma

  * Newly diagnosed disease
  * Stage II, III, or IV disease
* Measurable disease, defined as ≥ 1 lesion ≥ 1.5 cm in one diameter, as detected by CT scan or PET-CT scan (PET/CT fusion)
* CD20-positive disease
* No post-transplant lymphoproliferative disorder (PTLD)
* No CNS lymphoma or cerebrospinal fluid involvement with malignant lymphoma cells

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) OR direct bilirubin normal
* Alkaline phosphatase ≤ 3 times ULN (5 times ULN if direct liver involvement by lymphoma)
* AST ≤ 3 times ULN (5 times ULN if direct liver involvement by lymphoma)
* Creatinine ≤ 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective double-method contraception for ≥ 28 days before, during, and for ≥ 28 days after completion of study therapy
* Fertile male patients must use effective contraception during and for ≥ 28 days after completion of study therapy, even if they have had a successful vasectomy
* No blood, sperm, or semen donation during and for ≥ 28 days after completion of study therapy
* Willing to return to enrolling institution for follow-up
* Willing to provide blood samples for translational research purposes
* No comorbid systemic illness or other severe concurrent disease that, in the judgment of the investigator, would preclude study entry or significantly interfere with the proper assessment of safety and toxicity of the prescribed study regimen
* No known HIV positivity
* Not immunocompromised
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situation that would preclude compliance with study requirements
* No other active malignancy, except localized nonmelanotic skin cancer or any cancer that, in the judgment of the investigator, has been treated with curative intent and will not interfere with the study treatment plan and response assessment
* No myocardial infarction within the past 6 months
* No congestive heart failure requiring ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Ejection fraction ≥ 45% by MUGA or ECHO
* No history of life threatening or recurrent thrombosis/embolism (unless on anticoagulation therapy during study treatment)

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to ≥ 25% of the bone marrow
* No concurrent erythroid-stimulating agents (e.g., Procrit, Aranesp)
* No other concurrent treatment for lymphoma
* No concurrent radiotherapy, chemotherapy, or immunotherapy for another active malignancy
* Able to receive concurrent prophylactic anticoagulation therapy (e.g., low-dose aspirin [81 mg] daily or an alternative prophylaxis [e.g., warfarin or low molecular weight heparin])

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-08-25 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz S. Nowakowski, M.D., Study Chair — Mayo Clinic; Allison C. Rosenthal, D.O., Principal Investigator — Mayo Clinic; Candido E. Rivera, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Nowakowski GS, LaPlant B, Macon WR, Reeder CB, Foran JM, Nelson GD, Thompson CA, Rivera CE, Inwards DJ, Micallef IN, Johnston PB, Porrata LF, Ansell SM, Gascoyne RD, Habermann TM, Witzig TE. Lenalidomide combined with R-CHOP overcomes negative prognostic impact of non-germinal center B-cell phenotype in newly diagnosed diffuse large B-Cell lymphoma: a phase II study. J Clin Oncol. 2015 Jan 20;33(3):251-7. doi: 10.1200/JCO.2014.55.5714. Epub 2014 Aug 18. PMID 25135992

RESULTS

PARTICIPANT FLOW:
Groups:
- Ph 1, DL 1: Phase 1, Dose Level 1 lenalidomide 15 mg
- Ph1, DL 2: Phase 1, Dose Level 2 lenalidomide 20 mg
- Ph1, DL 3: Phase 1, Dose Level 3 lenalidomide 25 mg
- Ph II, DLBCL/Mixed: Phase 2, DLBCL/Mixed Dose Level 3 (accrued before 1/1/13)
- Ph II, Transformed/Composite: Phase 2, Transformed/Composite
- Ph II, Additional DLBCL: Phase 2, Additional DLBCL. Accrued after cutoff date
Period: Overall Study
Arm/Group | Ph 1, DL 1 | Ph1, DL 2 | Ph1, DL 3 | Ph II, DLBCL/Mixed | Ph II, Transformed/Composite | Ph II, Additional DLBCL
Started | 3 | 3 | 6 | 77 | 39 | 10
Completed | 3 | 3 | 5 | 59 | 33 | 0
Not Completed | 0 | 0 | 1 | 18 | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Ph 1, DL 1: Phase 1, Dose Level 1
- Ph1, DL 2: Phase 1, Dose Level 2
- Ph1, DL 3: Phase 1, Dose Level 3
- Total: Total of all reporting groups
Arm/Group | Ph 1, DL 1 | Ph1, DL 2 | Ph1, DL 3 | Ph II, DLBCL/Mixed | Ph II, Transformed/Composite | Ph II, Additional DLBCL | Total
Number analyzed (Participants) | 3 | 3 | 6 | 77 | 39 | 10 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (16.26) | 65.7 (14.36) | 70.2 (11.18) | 60.6 (15.99) | 64.7 (11.38) | 66.1 (13.10) | 62.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 29 | 18 | 4 | 56
  Male | 2 | 1 | 4 | 48 | 21 | 6 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 6 | 75 | 38 | 9 | 134
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 3 | 3 | 6 | 76 | 39 | 10 | 137
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Toxicity as Assessed by NCI CTCAE v3.0 (Phase I)
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 1, DL 1 | Ph1, DL 2 | Ph1, DL 3
Number analyzed (Participants) | 3 | 3 | 5
Participants
  Grade 3+ Adverse Event | 3 | 3 | 5
  Grade 4+ Adverse Event | 2 | 1 | 4
  Grade 3+ Hem Adverse Event | 3 | 3 | 5
  Grade 4+ Hem Adverse Event | 2 | 1 | 4
  Grade 3+ Non-Hem Adverse Event | 1 | 1 | 2

2. Primary Outcome: Event-free > Survival at 12 Months (Phase 2, DLBCL/Mixed Dose Level 3)
Description: Other Phase II Cohorts were not evaluable for event-free survival analysis.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ph II, DLBCL/Mixed
Number analyzed (Participants) | 64
Participants | 44

3. Primary Outcome: Progression-free > Survival at 24 Months (Phase 2, Transformed/Composite)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
  Other Phase II Cohorts were not evaluable for progression-free survival analysis.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ph II, Transformed/Composite
Number analyzed (Participants) | 33
Participants | 27

4. Secondary Outcome: Overall Response Rate
Time Frame: When all patients either have a CR or have completed observation.
Reporting Status: Not Posted

5. Secondary Outcome: Overall Complete Response Rate
Time Frame: When all patients either have a CR or have completed observation.
Reporting Status: Not Posted

6. Secondary Outcome: Event-free Survival
Time Frame: 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival
Time Frame: 5 years
Reporting Status: Not Posted

8. Secondary Outcome: Progression-free Survival
Time Frame: 5 years
Reporting Status: Not Posted

9. Secondary Outcome: Duration of Response
Time Frame: 5 years
Reporting Status: Not Posted

10. Secondary Outcome: Immune Function Before and After Treatment as Assessed by T-, B-, and NK-cell Quantification
Time Frame: 5 years
Reporting Status: Not Posted

11. Secondary Outcome: Correlation of Immune Function With Clinical Outcomes
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Ph 1, DL 1 | Ph1, DL 2 | Ph1, DL 3 | Ph II, DLBCL/Mixed | Ph II, Transformed/Composite | Ph II, Additional DLBCL
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 1/76 | 0/39 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 2/6 | 26/76 | 15/39 | 7/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 76/76 | 39/39 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph 1, DL 1 (N=3) | Ph1, DL 2 (N=3) | Ph1, DL 3 (N=6) | Ph II, DLBCL/Mixed (N=76) | Ph II, Transformed/Composite (N=39) | Ph II, Additional DLBCL (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (9) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Sepsis(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Skin infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 2 (3) | 1 (2) | 1 (1) | 8 (9) | 4 (4) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3) | 1 (3) | 0 (0) | 11 (18) | 4 (4) | 7 (10)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph 1, DL 1 (N=3) | Ph1, DL 2 (N=3) | Ph1, DL 3 (N=6) | Ph II, DLBCL/Mixed (N=76) | Ph II, Transformed/Composite (N=39) | Ph II, Additional DLBCL (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (5) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (22) | 3 (20) | 6 (40) | 75 (434) | 39 (260) | 10 (72)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 3 (5) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric mucositis (clin exam) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric mucositis (funct/sympt) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Mucositis oral (clin exam) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 10 (16) | 5 (5) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (9) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 20 (45) | 10 (26) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bladder infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Colitis, infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Kidney infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral nerve infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sepsis(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Sinusitis(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Skin infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tooth infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Upper respiratory infectn(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Vaginal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intraop. inj. - Colon (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 3 (10) | 3 (13) | 6 (27) | 74 (357) | 38 (200) | 10 (47)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 33 (174) | 3 (7)
Neutrophil count decreased (Investigations) | 3 (8) | 3 (10) | 6 (25) | 71 (318) | 36 (176) | 9 (36)
Platelet count decreased (Investigations) | 3 (15) | 3 (14) | 6 (27) | 70 (318) | 38 (196) | 9 (50)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (10) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 1 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 3 (7) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (3) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (5) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 2 (2) | 1 (3) | 9 (19) | 4 (11) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (5) | 2 (9) | 3 (13) | 44 (178) | 27 (102) | 4 (17)
Hand-and-foot syndrome/reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT00670358/Prot_SAP_000.pdf